CLINICAL TRIAL: NCT05165615
Title: Comparison of the Two Different Closed-loop Hybrid Systems - AndroidAPS and Control-IQ in Patients With Type 1 Diabetes
Brief Title: Android Artificial Pancreas System (Android APS) Versus Control-IQ
Acronym: CODIAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Soupal, MD, Principal Investigator, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CODIAC
Record Dates: First submitted 2021-11-23; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitoring; Insulin Pump; Closed-loop hybrid system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AndroidAPS versus Control-IQ (Experimental): Patients with use of the Control-IQ system (closed-loop hybrid system) and previous users of AndroidAPS (closed-loop hybrid system)
  Interventions: Device: Insulin Pump t:slim X2 with Control-IQ technology

INTERVENTIONS:
Device: Insulin Pump t:slim X2 with Control-IQ technology — Usage of Insulin pump t:slim X2 with Control-IQ technology in previous users of AndroidAPS
  Other Names: Continuous Glucose Monitoring Dexcom G6 system

SUMMARY:
The aim of the investigator's study is to compare two different closed loop hybrid systems - certified Control-IQ and noncertified AndroidAPS in adult patients with Type 1 Diabetes (T1D), who had been using AndroidAPS previously from their own decision, during 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed >2 years
* ≥ 18 years old
* written informed consent prior to starting study related activity
* previous user of AndroidAPS at least for 3 months

Exclusion Criteria:

* severe noncompliance
* lactation, pregnancy, intending to become pregnant during study
* use of medication with effects on carbohydrate metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in target ranges | Up to 28 weeks
  3.9-10.0 mmol/L (70-180 mg/dl)

SECONDARY OUTCOMES:
Percentage of time in hypoglycemic ranges | Up to 28 weeks
  <3.9 mmol/L (70 mg/dl) and <3.0 mmol/L (54 mg/dl)
Percentage of time in hyperglycemic ranges | Up to 28 weeks
  >10.0 mmol/L (180 mg/dl) and >13.9 mmol/L (250 mg/dl)
Changes in glycemic variability | Up to 28 weeks
  Expressed as the coefficient of variation
Incidence of severe hypoglycaemia | Up to 28 weeks
  Requiring third-party assistance to treat
Changes in glycated haemoglobin (HbA1c) | Up to 28 weeks
  Differences between HbA1c values in the initial period and after follow-up
Hypoglycemia Attitudes and Behavior Scale (HABS) | Up to 28 weeks
  This validated questionnaire contains in total 14 questions that highlights two critical dimensions of hypoglycemia-related concerns (anxiety and avoidance) and one positive dimension (confidence). 14 items use Likert scales from 1 to 5, total score from 14 to 70, the higher total score means worse outcome.
Diabetes Distress Scale (DDS) | Up to 28 weeks
  This validated questionnaire assess diabetes-related emotional stress. This 17-item tool uses the Likert scales from 1 to 6. Total score is from 17 to 102, while higher total score means worse outcome.
The 5-item World Health Organization well-being index (WHO-5 index) | Up to 28 weeks
  This validated questionnaire contains in total 5 questions with Likert scales from 5 to 0. Total score is multiplied by 4 to give a final score ranging from 0 to 100, higher score denote higher quality of life (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Soupal, Principal Investigator — Charles University, Prague
Locations (1):
- 3rd Department of Internal Medicine, 1st Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hajos TR, Pouwer F, Skovlund SE, Den Oudsten BL, Geelhoed-Duijvestijn PH, Tack CJ, Snoek FJ. Psychometric and screening properties of the WHO-5 well-being index in adult outpatients with Type 1 or Type 2 diabetes mellitus. Diabet Med. 2013 Feb;30(2):e63-9. doi: 10.1111/dme.12040. PMID 23072401
- [Background] Fisher L, Hessler DM, Polonsky WH, Mullan J. When is diabetes distress clinically meaningful?: establishing cut points for the Diabetes Distress Scale. Diabetes Care. 2012 Feb;35(2):259-64. doi: 10.2337/dc11-1572. Epub 2012 Jan 6. PMID 22228744
- [Background] Polonsky WH, Fisher L, Hessler D, Liu J, Fan L, McAuliffe-Fogarty AH. Worries and concerns about hypoglycemia in adults with type 1 diabetes: An examination of the reliability and validity of the Hypoglycemic Attitudes and Behavior Scale (HABS). J Diabetes Complications. 2020 Jul;34(7):107606. doi: 10.1016/j.jdiacomp.2020.107606. Epub 2020 Apr 23. PMID 32354623
- [Background] Soupal J, Petruzelkova L, Grunberger G, Haskova A, Flekac M, Matoulek M, Mikes O, Pelcl T, Skrha J Jr, Horova E, Skrha J, Parkin CG, Svacina S, Prazny M. Glycemic Outcomes in Adults With T1D Are Impacted More by Continuous Glucose Monitoring Than by Insulin Delivery Method: 3 Years of Follow-Up From the COMISAIR Study. Diabetes Care. 2020 Jan;43(1):37-43. doi: 10.2337/dc19-0888. Epub 2019 Sep 17. PMID 31530663
- [Background] Soupal J, Petruzelkova L, Flekac M, Pelcl T, Matoulek M, Dankova M, Skrha J, Svacina S, Prazny M. Comparison of Different Treatment Modalities for Type 1 Diabetes, Including Sensor-Augmented Insulin Regimens, in 52 Weeks of Follow-Up: A COMISAIR Study. Diabetes Technol Ther. 2016 Sep;18(9):532-8. doi: 10.1089/dia.2016.0171. Epub 2016 Aug 2. PMID 27482825
- [Background] Haskova A, Radovnicka L, Petruzelkova L, Parkin CG, Grunberger G, Horova E, Navratilova V, Kade O, Matoulek M, Prazny M, Soupal J. Real-time CGM Is Superior to Flash Glucose Monitoring for Glucose Control in Type 1 Diabetes: The CORRIDA Randomized Controlled Trial. Diabetes Care. 2020 Nov;43(11):2744-2750. doi: 10.2337/dc20-0112. Epub 2020 Aug 28. PMID 32859607